CLINICAL TRIAL: NCT07260448
Title: Immediate Effects of Paraffin Wax Therapy on the Forearm and Hand Muscles' Stiffness and Pain in Patients With Carpal Tunnel Syndrome: A Randomised Controlled Trial
Brief Title: Immediate Effects of Paraffin Wax Therapy on Forearm and Hand Muscle Stiffness and Pain in Carpal Tunnel Syndrome
Acronym: Paraffin-CTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Amasya University (Other); Bangor University (Other)
Responsible Party: Principal Investigator, esedullah akaras, Dr., Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETU-P-WAX-CTS Trial
Record Dates: First submitted 2025-11-19; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome (CTS); Muscle Stiffness
Keywords: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants with carpal tunnel syndrome will be randomly assigned (1:1) to paraffin wax therapy or a control group; muscle stiffness and pain will be assessed immediately before and after the session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paraffin Wax Therapy (Experimental): Participants receive a single session of paraffin wax therapy to the affected hand and forearm. Muscle stiffness and pain are assessed immediately before and after the session.
  Interventions: Other: Paraffin Wax Therapy; Other: Rest Period (No Treatment)
- Rest / Control (Other): Participants rest quietly for 20 minutes in a comfortable position with the forearm supported, without receiving paraffin wax or any other physical/thermal modality. Muscle stiffness and pain are assessed at the same time points as in the experimental arm.
  Interventions: Other: Paraffin Wax Therapy; Other: Rest Period (No Treatment)

INTERVENTIONS:
Other: Paraffin Wax Therapy — Participants in the experimental arm receive paraffin wax therapy to the affected hand and forearm. Melted paraffin is maintained at approximately 42-44 °C. Using a brush-on technique, 10 consecutive layers of wax are applied, and the limb is then covered with a plastic glove and towel to retain heat. The participant remains seated with the forearm supported in a relaxed position for 20 minutes. Muscle stiffness (MyotonPro) and pain are measured immediately before and within 5 minutes after the session.
Other: Rest Period (No Treatment) — Participants in the control arm rest quietly for 20 minutes in a comfortable seated or supine position with the forearm supported. No thermal, manual or exercise-based treatment is provided during this period. Muscle stiffness (MyotonPro) and pain are measured immediately before and within 5 minutes after the rest period, using the same procedures and time points as in the experimental arm.

SUMMARY:
This randomized controlled trial aims to investigate the immediate effects of paraffin wax therapy on muscle stiffness and pain among patients diagnosed with Carpal Tunnel Syndrome (CTS). The intervention involves immersing the hand and forearm in paraffin wax at 42-44 °C for 20 minutes. Stiffness will be measured using the MyotonPro device, and pain will be evaluated using standard visual scales.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy of the upper limb and may alter the passive mechanical properties of forearm and hand muscles, contributing to pain and functional limitation. Handheld devices such as MyotonPro allow non-invasive, point-of-care assessment of muscle stiffness, elasticity and viscoelastic behaviour in clinical settings. Paraffin wax therapy is widely used as a superficial heat modality in hand rehabilitation and has been shown to reduce pain and improve function in various hand conditions, but its immediate effects on objectively measured muscle stiffness in CTS remain unclear. This parallel-group randomised controlled trial will examine the immediate effects of a single paraffin wax session on muscle stiffness and pain in adults with CTS. Physically active adults aged 18-65 years with clinically diagnosed CTS will be recruited from university-based facilities in Erzurum, Türkiye, and randomly allocated (1:1) to paraffin wax therapy or a control condition. A priori power analysis indicated that a total sample of 24 participants (12 per group) would provide adequate power to detect between-group differences in pre- to post-intervention change. Mechanical properties of selected forearm and hand muscles (e.g. APB, FDS, ECRB, FCU) will be assessed using MyotonPro immediately before and after the intervention. In the intervention group, the affected hand and forearm will receive 20 minutes of paraffin wax therapy at approximately 42-44 °C using a standardised brush-on technique and safety checks for skin integrity and temperature. Pain intensity in the affected region will be recorded pre- and post-session using a validated numeric rating or similar pain scale. The primary outcome is the between-group difference in immediate change in MyotonPro stiffness parameters, with secondary outcomes including change in pain and exploratory relationships between changes in stiffness and pain. Mixed model repeated measures ANOVA will be used to compare pre- to post-intervention changes between groups. Findings from this study may help clarify the short-term neuromuscular and symptomatic effects of paraffin wax therapy in CTS and inform future rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed carpal tunnel syndrome.
* Age between 18 and 65 years.
* Apparently healthy, without a known chronic systemic disease (other than CTS).
* No history of other chronic musculoskeletal or neurological disorders.

Exclusion Criteria:

* Previous surgery on the affected wrist or hand.
* Systemic conditions affecting nerve function (e.g., diabetes mellitus, thyroid disease)
* Cardiovascular disease or uncontrolled hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Change in muscle stiffness parameters | Immediately before the intervention and within 5 minutes after completion of the 20-minute paraffin/rest session (same visit)
  Change in MyotonPro-derived muscle stiffness (Newton per metre) of selected forearm and hand muscles (adductor pollicis brevis, flexor digitorum superficialis, extensor carpi radialis brevis, flexor carpi ulnaris ). For each site, three consecutive impulses separated by at least 10 seconds will be averaged. The primary comparison is the between-group difference (paraffin vs rest) in pre- to post-session change scores.

SECONDARY OUTCOMES:
Change in pain intensity | Immediately before the intervention and within 5 minutes after completion of the 20-minute paraffin/rest session (same visit).
  Change in self-reported pain intensity in the affected hand/forearm, assessed using a numeric rating scale (0 = no pain, 10 = worst imaginable pain). The main comparison is between-group difference in pre- to post-session change scores. Pain assessments are performed at the same time points as MyotonPro measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Şehir Hastanesi, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this trial. Summary results and aggregate data will be disseminated through peer-reviewed publications and conference presentations.